CLINICAL TRIAL: NCT00550160
Title: The Clinical Impact of Seasonal Intermittent Preventive Treatment (IPT) and Home Management of Malaria (HMM) Using AQ+AS in Ghanaian Children Under 5 Years of Age - a Cluster Randomised Placebo Controlled Trial.
Brief Title: The Synergistic Effects of Home-management and Intermittent Preventive Treatment of Malaria in Children
Acronym: KNUST-COMDIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kwame Nkrumah University of Science and Technology (Other)
Collaborators: Department for International Development, United Kingdom (Other Government); Malaria Consortium, UK (Network); Center for International Health and Development (Other)
Responsible Party: Principal Investigator, Dr. Harry Tagbor, Dr, Kwame Nkrumah University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CKNT_1
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): The Home Management of Malaria (HMM) is a strategy aimed at improving access to prompt and effective antimalarial treatment of all fevers in children under 5 years. Community Drug Distributors (CDD) have been trained and equipped for this task.
  Interventions: Drug: Amodiaquine plus Artesunate co-administration
- 2 (Experimental): An Intermittent Preventive Treatment (IPTc) schedule for asymptomatic pre-school children during high malaria transmission seasons alongside an ongoing Home Management of Malaria programme
  Interventions: Drug: Amodiaquine plus Artesunate co-administration

INTERVENTIONS:
Drug: Amodiaquine plus Artesunate co-administration — Under the Home Management of Malaria (HMM) strategy the Community Drug Distributors (CDD) will treat all children under 5 years presented to them with measured fever or a history of fever with AQ plus AS co-administered. Children under 12 months receive 75mg of AQ co-administered with 25mg of AS daily for three days. Children who are 12 to 59 months old receive 150mg of AQ and 50mg of AS co-administered daily for three days.
  Asymptomatic children under 5 years in the Intermittent Preventive Treatment (IPTc) clusters will receive additional AQ plus AS co-administered during high malaria transmission season. Those under 12 months will receive 75mg of AQ co-administered with 25mg of AS daily for three days; and children who are 12 to 59 months old receive 150mg of AQ and 50mg of AS co-administered daily for three days.

SUMMARY:
This cluster randomised trial is proposed to assess the clinical impact of adding a seasonal intermittent preventive treatment (IPTc) schedule for children aged 3 -59 months to a home management of malaria (HMM) programme using AQ+AS in Ghana. The study will be conducted in the Kwaso sub district of the Ejisu-Juaben district of Ghana in which 6 communities will be randomised to implement an IPTc schedule alongside the HMM programme or HMM programme alone.

The study will run in three phases; a preparatory phase to set up and obtain baseline morbidity data from a cross-sectional survey; an intervention phase and a post intervention phase of cross-sectional survey and data evaluation and dissemination. A cohort of 546 study children randomly selected will receive three full treatment courses of AS+AQ intermittently during the April - Nov 2007 transmission season. Community-based drug distributors (CDDs) will administer all courses of IPTc. The first dose of each course will be directly observed by the CDDs who will educate mothers or caregivers to administer subsequent doses appropriately at home. Follow up visits to homes will be done by CDDs and field supervisors to ascertain adherence and to monitor adverse drug events. The incidence of clinical malaria and other secondary outcomes will be compared with those of another cohort of 546 study children who will not receive IPTc but may be treated under the HMM strategy alone with AS+AQ when necessary during the observation period.

ELIGIBILITY:
Inclusion Criteria:

* A child in the study cohort will be eligible to receive a course of IPTc (active or placebo) if the child has NO fever (a temperature of 37•5o C or above) or history of fever in the last 24 hours. However, fever is only a temporary exclusion criterion. If a child has fever when he/she is due for an IPTc course, treatment will be given for the fever and the IPTc course given one month after the fever has subsided. This interval between treatment of fever episodes and administration of an IPTc course is proposed in order to minimise the risk of overdosing since the same drug is used for both HMM and IPTc.

Exclusion Criteria:

* A child in the study cohort will not be eligible to receive a course of IPTc if:

  * The child has a clinical condition that may be classified as severe according to IMCI guidelines.
  * The child is known to suffer from chronic disease(s) e.g. sickle cell disease that might adversely affect the interpretation of study results.
  * The mother/caregiver withdraws consent.

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1490 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Incidence rate of clinical episodes of malaria per child per year | One year

SECONDARY OUTCOMES:
Prevalence of peripheral parasitaemia | One year
Prevalence of anaemia | One year
Parasite density (geometric means) | One year
Proportions adhering to strategies | One year
Incidence of adverse drug effects within 7 days after intervention | One year

CONTACTS AND LOCATIONS:
Overall Officials: Harry Tagbor, DrPH, Principal Investigator — Department of Community Health, School of Medical Science, Kwame Nkrumah University of Science & Technology; Edmund Browne, PhD, Principal Investigator — Department of Community Health, School of Medical Sciences, Kwame Nkrumah University of Science & Technology; Helen Counihan, PhD, Principal Investigator — Malaria Consortium, UK; Sylvia Meek, PhD, Principal Investigator — Malaria Consortium, UK
Locations (1):
- District Health Administration, Ejisu, Ashanti Region, Ghana